CLINICAL TRIAL: NCT04855929
Title: ANV419 First in Human Study Phase 1: Open-label, Dose Escalation Study of ANV419 As Single Agent and in Combination with Ipilimumab in Patients with Relapsed/Refractory Advanced Solid Tumors
Brief Title: A Study Evaluating Safety and Therapeutic Activity of ANV419 in Patients with Advanced Cancer.
Acronym: ANV419-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anaveon AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANV419-001
Record Dates: First submitted 2021-04-15; First posted 2021-04-22 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor; Adult Disease; Lung Cancer
Keywords: IL-2; ANV419; Cancer; Relapsed; Refractory; Ipilimumab
MeSH Terms: conditions — Disease; Lung Neoplasms; Neoplasms; Recurrence | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ANV419 single agent (Experimental)
  Interventions: Drug: ANV419
- Ipilimumab + ANV419 (Experimental)
  Interventions: Drug: ANV419; Drug: Ipilimumab

INTERVENTIONS:
Drug: ANV419 — ANV419 administered by intravenous (IV) infusion
Drug: Ipilimumab — Ipilimumab administered by intravenous (IV) infusion
  Arms: Ipilimumab + ANV419

SUMMARY:
The purpose of this study is to test the safety and efficacy of ANV419 (single agent) and in combination with ipilimumab in patients with relapsed/refractory advanced solid tumors.

DETAILED DESCRIPTION:
The purpose of this First-in-Human, open-label, dose escalation study is to assess the initial safety and efficacy profile of ANV419 intravenous infusion alone and in combination with ipilimumab in patients with advanced solid tumours. It will evaluate the safety and tolerability of ANV419 alone and in combination with ipilimumab and, the safest and best dose of ANV419 when used alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the patient or legal guardian to understand the purpose of the study, provide signed and dated informed consent from the patient prior to performing any protocol-related procedures (including Screening evaluations), and be able and willing to comply with the study procedures.
* Male or female aged ≥ 18 years.
* Advanced solid tumors with evidence of progressive disease as per RECIST no longer than 3 months before Informed Consent form (ICF) signature, without any subsequent curative intent treatment.
* Parts A and B only: Histologically confirmed relapsed/refractory advanced solid tumor, progressing after at least one line of treatment for advanced or metastatic disease
* Part C only: Previously treated advanced NSCLC without a driver mutation who have progressed after first line standard chemo-immunotherapy: Patients must have measurable disease using RECIST v1.1, A maximum of 1 line of therapy is permitted, Patients with high expression of PD-L1 which were treated with first line checkpoint inhibitor monotherapy may have received a maximum of 2 lines of therapy
* Part D only: Histologically confirmed relapsed/refractory advanced solid tumors progressing after at least one line of treatment for advanced disease. Patients with NSCLC who do not meet inclusion criteria for Part C, are eligible for Part D
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Adequate pulmonary, cardiovascular, hematological, liver and renal function, per Investigator judgment.
* All acute toxic effects, of any prior anticancer therapy (e.g., radiotherapy, chemotherapy, or surgical procedures) must have resolved to CTCAE v5.0 grade ≤1 (except alopecia [any grade] or fatigue [up to grade 2 allowed]).
* Negative serum pregnancy test at screening and a negative (urine or serum) pregnancy test within 7 days prior to study day 1 in women of childbearing potential and women <12 months after menopause.
* Women who are not postmenopausal and who have not undergone surgical sterilization: must agree to use highly effective methods of contraception during the treatment period and until 6 months after the last dose of study treatment. They must also agree to not donate eggs (ova, oocytes) during the same timeframe.
* All men with childbearing potential partners must agree to use highly effective methods of contraception and barrier contraception (condom) during the treatment period and for 6 months after the last dose of study treatment. They must also agree to not donate sperm during the same timeframe.
* Availability and willingness of patients to obtain a baseline and on treatment biopsy of the tumor. Available archived biopsies (frozen or formalin fixed) may serve as baseline specimens, in patients who have residual tumor masses which can only be accessed with significant risk

Exclusion Criteria:

* Carcinomatous meningitis and/or symptomatic central nervous system (CNS) metastases. Definitively treated CNS metastases (e.g., radiotherapy) stable for at least 6 weeks prior to Day 1 of study drug administration are acceptable.
* Participants with an active second malignancy. Patients with precancerous lesions, concomitant early stages of prostate or breast cancer not requiring active treatment (past conditions currently resolved > 3 years prior to Screening are also acceptable), and squamous cell carcinoma of the skin not requiring systemic treatment are acceptable.
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including uncontrolled diabetes mellitus, history of relevant pulmonary disorders, (e.g., severe bronchospasm, obstructive pulmonary disease), hyperthyroidism due to thyroiditis and known autoimmune diseases or other disease with ongoing fibrosis. Stable vitiligo, autoimmune thyroiditis, and preexisting treated type 1 diabetes are acceptable and are not exclusion criteria.
* Significant cardiovascular/cerebrovascular disease, including myocardial infarction or transient ischemic attack (TIA) within 6 months prior to Day 1 of study drug administration.
* Active infections, or uncontrolled infection requiring systemic antibiotics within one week (7 days) preceding Day 1 of treatment
* Hemoglobin (Hb) <9 g/dL, transfusion of red blood cells allowed to reach threshold target.
* Neutrophils <1500 /mm3.
* Platelets <100'000/mm3.
* Liver: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5xULN, if due to liver metastasis or primary liver cancer, AST or ALT >5x ULN.
* Total bilirubin > upper limit of normal (ULN) (in documented Gilbert's syndrome, direct bilirubin > ULN).
* International normalized ratio (INR) >1.5xULN.
* Serum creatinine > ULN and estimated creatinine clearance < 50 mL/min using the Cockcroft-Gault formula.
* Confirmed replicating human immunodeficiency virus (HIV) or confirmed active (replicative) hepatitis B virus or hepatitis C virus infection. Patients with treated non-replicative disease are acceptable.
* Evidence of hepatic cirrhosis with Child-Pugh score C.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding > Grade 2 that give reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug.
* Major surgery or significant traumatic injury <28 days prior to the first ANV419 infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment.
* Severe altered mental status.
* Pregnant or breastfeeding women.
* Known hypersensitivity to any of the components of ANV419 or its formulation.
* Concurrent therapy with any other investigational drug within one month prior to Day 1 of study drug administration.
* Active untreated immune-related endocrinopathies untreatable with replacement. Prior immune related toxicities > Grade 3 after treatment with immunostimulatory drugs (e.g., colitis, neuropathy) that have not completely resolved.
* Chronic treatment with systemic immunosuppressive medications above 10 mg/day prednisolone equivalent for any reason.

Additional exclusion criteria for Part D:

* Experienced unacceptable drug-related toxicity with prior ipilimumab treatment (defined as toxicities that required second line immunosuppression, ie, not controlled by steroids alone)
* Received ipilimumab within 6 months prior to cycle 1 day 1.
* Known hypersensitivity to ipilimumab or any of its excipients
* Patients with active autoimmune disease or a history of autoimmune disease (other than vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism),
* Symptomatic interstitial lung disease
* Concomitant use of therapeutic anti-coagulation (e.g.to treat pulmonary embolus or deep vein thrombosis). Prophylactic anti-coagulation is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Monotherapy: Number of Dose-Limiting Toxicities (DLTs) | Day 1 to Day 14
Combination: Number of Dose-Limiting Toxicities (DLTs) | Day 1 to Day 21
Monotherapy: Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to 12 months
Combination: Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to 12 months
Monotherapy: Recommended Phase 2 Dose | Day 1 to Day 28
Combination: Recommended Phase 2 Dose | Day 1 to Day 28

SECONDARY OUTCOMES:
Objective response rate (ORR) assessed by RECIST v1.1 for solid tumors | Day 1 up to 12 months
Plasma concentration of ANV419 in blood | Day 1 up to 12 months
Impact of ANV419 on the expression of markers of PBMC lineage in blood | Day 1 up to 12 months
Levels of specific anti-ANV419 antibodies in blood | Day 1 up to 12 months
Disease control according to RECIST v1.1 | Day 1 up to 12 months
Progression-free survival (PFS) according to RECIST v1.1 | Day 1 up to 12 months
Duration of response (DOR) according to RECIST v1.1 | Day 1 up to 12 months
Overall survival (OS) | Day 1 up to 12 months
Quality of life assessed with European Quality of Life Five Dimensions (EQ-5D-5L) | Day 1 up to 12 months
Quality of life assessed with European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Day 1 up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Gasal, MD, Study Director — Anaveon AG
Locations (5):
- Spain (2):
  - Hospital Vall d'Hebrón, Barcelona
  - START Madrid, Hospital Universitario HM Sanchinarro, Madrid
- Switzerland (2):
  - University Hospital Basel, Basel
  - Cantonal Hospital St.Gallen, Sankt Gallen
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joerger M, Calvo E, Laubli H, Lopez J, Alonso G, Corral de la Fuente E, Hess D, Konig D, Sanchez Perez V, Bucher C, Jethwa S, Garralda E. Phase 1 first-in-human dose-escalation study of ANV419 in patients with relapsed/refractory advanced solid tumors. J Immunother Cancer. 2023 Nov 21;11(11):e007784. doi: 10.1136/jitc-2023-007784. PMID 38243906